CLINICAL TRIAL: NCT00096902
Title: Non-Pharmacologic Therapy for Neurocardiogenic Syncope
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050024; 05-N-0024
Record Dates: First submitted 2004-11-16; First posted 2004-11-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-09-11

CONDITIONS: Syncope
Keywords: Orthostatic Intolerance; Hypnosis; Cold Pressor; Isometric Exercise; Behavior; Neurocardiogenic Syncope
MeSH Terms: conditions — Syncope; Orthostatic Intolerance; Behavior; Syncope, Vasovagal

INTERVENTIONS:
Procedure: Tilt table test

SUMMARY:
This study will examine whether certain procedures that do not involve the use of medications can reduce symptoms of neurocardiogenic syncope (SIN-ku-pe), or a condition involving recurrent fainting. This condition is also known as vasovagal syncope or neurally mediated hypotension. Neurocardiogenic syncope is a disorder of the autonomic nervous system, which controls automatic body functions such as blood pressure, heart rate, and sweating. That system can be affected by medications, conditions of the mind or body, and by a person's surroundings. Researchers in this study wish to learn whether hypnosis, hand exercises, education, or diary keeping can affect the autonomic nervous system and improve symptoms of neurocardiogenic syncope.

Patients age 18 or older who have neurocardiogenic syncope may be eligible for this study. Those who have a medical illness making it unsafe to participate, who cannot discontinue certain medications, or who are pregnant are not eligible. Patients will undergo a medical history and physical examination, complete a questionnaire, and experience Valsalva and tilt table tests. These tests will take about 5 hours during 1 to 2 days.

The Valsalva test evaluates some of the reflexes of autonomic nervous system. Patients will lie flat on a padded table and have sensors placed on the body, to measure blood pressure, breathing rate, and other functions. They will blow into a sterile tube for 12 seconds while the body's responses are measured. The procedure may need to be repeated several times. During the test, an intravenous tube, guided by a needle, will be placed in the patient's arm. The tube will be used to collect samples of blood (less than 7 tablespoons) to measure chemicals such as adrenaline. For the tilt table test, a patient will lie on a padded, motorized table and have sensors placed on the body. Velcro straps will be placed around the patient's body to help hold him/her on the table. Then the table will tilt the patient from a flat position to an upright one in about 10 seconds. The patient will stay upright for 45 minutes while symptoms are monitored, measurements are taken, and blood samples are collected through the intravenous tube. Then the table will be returned to the flat position. If the patient faints or is about to faint, or if he or she has an unsafe heart rhythm before the 45 minutes is over, the test will be stopped and the table will be returned to the flat position. Symptoms will be treated as needed.

Patients who qualify for further study will then become familiar with hypnosis and be evaluated for their natural ability for experiencing it. A professionally trained doctor will guide patients into a hypnotic state, and patients will be asked to respond to various suggestions. They will be videotaped, an activity that will require a separate consent form. Following these procedures, patients will be assigned to one of the four groups in this study. Those in the hypnosis group will have weekly sessions for 6 weeks, with each session lasting about 1-1/2 hours. The education group will meet a study investigator for learning about syncope and the autonomic nervous system, with each session lasting about 1-1/2 hours once a week for 6 weeks. The hand exercise group will be taught certain hand exercises to perform, at home and as instructed, for 6 weeks. The diary group will receive instructions on keeping a diary pertaining to their condition, at home, for 6 weeks. After 6 weeks, patients will return for an evaluation to include completion of questionnaires and another tilt table test and blood collection by intravenous tube. This entire study will take about 8 weeks. There may be direct benefits from participating in this study. The experimental procedures may help patients' neurocardiogenic syncope.

After completing this study, patients will be offered any or all of the experimental procedures tested in this study upon their request and at the discretion of the principal investigator. For example, a patient who is assigned to the diary group may be offered hypnosis, education, and hand exercise instruction after completion of the study.

DETAILED DESCRIPTION:
Objective: The objective of this protocol is to test the efficacy of non-pharmacologic interventions for recurrent neurocardiogenic syncope. Specifically, the interventions tested in this study are hypnosis, patient education, hand exercises, and diary-keeping.

Study Population: Subjects are patients ages 18 years or older with recurrent neurocardiogenic syncope or presyncope.

Design: Patients who have a positive screening tilt table test are assigned to one of four groups: hypnosis, patient education, hand exercises, or diary-keeping. Following 6 weeks of outpatient intervention, all patients undergo repeat tilt table testing to complete the study.

Outcome Measures: The primary outcome measure is occurrence of syncope or presyncope during upright tilt table testing. Secondary measures are hemodynamic and neurochemical parameters during upright tilt table testing, and quality of life measures including recurrence of outpatient syncopal episodes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects are patients referred for neurocardiogenic syncope or presyncope, with or without postural tachycardia syndrome (POTS). Patients enter the trial after positive tilt table testing during the screening evaluation. Participation is offered to individuals 18 years old or older, independently of gender, race, advanced age, ethnicity, religion, or any other demographic or sociopolitical classifications.

EXCLUSION CRITERIA:

Minors younger than 18 years old are excluded. Advanced age is not an exclusion criterion.

Patients who have certain illnesses that would interfere or be contraindicated with the interventions or procedures in this study are excluded. These include significant coronary artery disease, psychosis, or psychotic depression.

A candidate is excluded if the subject is unwilling to experience hypnosis or to have hypnosis sessions recorded; holds religious or other beliefs that would prevent engagement in hypnosis; is not fluent in spoken English; or has physical or other disabilities that prevent adequate participation in hypnotic susceptibility testing.

Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements must be discontinued before enrollment in the study. For many herbal medicines or dietary supplements, the mechanisms of action and therefore the possible effects on the experimental results are unknown. In cases where the subjects wish to continue their herbal medicines or dietary supplements while on study, and search of the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate.

A candidate is excluded if clinical considerations require that the patient continue treatment with a drug likely to interfere with the scientific results. Patients who cannot discontinue medications in the following categories are excluded: certain anti-hypertensives including beta-blockers, anticoagulants, tricyclic antidepressants, barbiturates, and acetaminophen. Patients unable to discontinue nicotine, caffeine, or alcohol for 24 hours prior to tilt table testing are excluded. Patients with chronic alcohol intake are excluded. Patients are not to discontinue any medications before the patient or the patient's doctor discusses this with the Principal Investigator, Accountable Investigator, an Associate Investigator, or Research Nurse. If it is decided that discontinuing medications would be unsafe, then the patient is excluded.

Patients who pose technical difficulties regarding the testing procedures are excluded.

A candidate is excluded if, in the judgment of the Principal Investigator, Accountable Investigator, or Clinical Director, protocol participation would place the subject at substantially increased acute medical risk, or if the medical risk outweighs the potential scientific benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-11-08; Study Completion 2006-09-11

PRIMARY OUTCOMES:
Occurrence of syncope or presyncope during upright tilt table testing.

SECONDARY OUTCOMES:
Hemodynamic and neurochemical parameters during upright tile table testing, and quality of life measures including recurrence of outpatient syncopal episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldstein DS, Holmes C, Frank SM, Naqibuddin M, Dendi R, Snader S, Calkins H. Sympathoadrenal imbalance before neurocardiogenic syncope. Am J Cardiol. 2003 Jan 1;91(1):53-8. doi: 10.1016/s0002-9149(02)02997-1. PMID 12505571